CLINICAL TRIAL: NCT06357962
Title: Clinical Trial With Two Branches to Study the Effect of Semi-permanent Acupuncture at Specific Acupuncture Points on Reducing the Number of Inductions During Labor in Women at Low or Moderate Risk
Brief Title: Semi-permanent Acupuncture Effect on Cervical Ripening
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources to continue the study
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CSAPG-40
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy Complications
Keywords: Cervical Ripening; Acupuncture Therapy
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): This group will receive sessions the study intervention (semi-permanent acupuncture)
  Interventions: Other: Semi-permanent acupuncture
- Control (Sham Comparator): This group will receive a sham treatment of semi-permanent acupuncture
  Interventions: Other: Sham of semi-permanent acupuncture

INTERVENTIONS:
Other: Semi-permanent acupuncture — These are sessions that last approximately one hour. The selection of points will be based on the energy diagnosis made during the first visit. In some cases, a point may be changed depending on progress. During the session, an interrogation will be conducted to assess symptoms and signs of the condition, and to evaluate if there have been any adverse reactions to the previous session. At the end of the visit, semi-permanent acupuncture will be applied to the selected points.
  Arms: Acupuncture
Other: Sham of semi-permanent acupuncture — A simulated semi-permanent acupuncture session will be conducted, consisting of specific placebo materials without needles and without stimulation for a few minutes. These points will not correspond to any acupuncture point and will be located on the hands, feet, and back. Stickers without pins will be applied, but never in critical points related to contraction stimulation or cervical ripening.
  Arms: Control

SUMMARY:
Cervical ripening is a medical treatment that can cause physical or emotional discomfort in pregnant women and is not without risks. This is a pilot study to assess feasibility and calculate the number of participants necessary for a complete clinical trial. The aim is to evaluate whether acupuncture can reduce the need for treatment (cervical ripening) in pregnant women at low or intermediate risk. Participants will be divided into two groups: one group will receive acupuncture, and the other will receive a simulated treatment of acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated delivery at the study center.
* Ability to collaborate in necessary evaluations.
* Legal capacity to provide informed consent.
* Signature of the informed consent for inclusion in the study, by oneself.

Exclusion Criteria:

* Pregnancy with high or very high risk as described by the Pregnancy and Childbirth Monitoring Protocols of the Department of Health of Catalonia
* History of cesarean delivery.
* Language barrier preventing collaboration in study procedures.
* Cognitive or affective pathology limiting the ability to collaborate with study procedures.
* Participation in another clinical trial involving an experimental intervention during the period of this trial and/or establishing a visit frequency incompatible with this trial.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The participants will be pregnant women
Enrollment: 8 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
Pharmacological induction | Birth date
  Percentage of pregnant women who have undergone pharmacological induction to initiate labor.

SECONDARY OUTCOMES:
Change on score of Bishop scale | Birth date
  Change from the initial obstetric assessment (weeks 36 to 38 of gestation) to the day of admission for delivery in the total score of the Bishop scale
Onset of spontaneous labor | Birth date
  Time in days until the onset of spontaneous labor from the first follow-up visit.
Duration of induction period Duration of the induction period Duration of the induction period Duration of the induction period | Birth date
  Time in hours from the administration of medication for induction to the onset of labor.
Duration of labor period | Birth date
  Time in hours of labor period
Satisfaction of pregnants | Birth date
  Degree of satisfaction with the care provided, measured by conducting the Birth Satisfaction Scale Revised survey

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Villena, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedes i Garraf, Vilafranca del Penedès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.